CLINICAL TRIAL: NCT07206186
Title: Music Listening During Anesthesia Induction and Emergence: Assessing Its Role in Enhancing Patient Comfort
Brief Title: Effect of Music on Patient Comfort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marion Wiegele, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1166/2025
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Anxiety
Keywords: Perioperative Anxiety; Music; Music intervention; State Trait Anxiety Inventory (STAI); NASA Task Load Index; Anesthesia; Patient Comfort
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Masking Description: Due to the study design (i.e. listening to music over a speaker), masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): After randomization, the intervention group will be asked which type of music they would like to listen to during anesthesia induction and emergence. Upon arrival in the operating room, the selected music will be played from a wireless speaker at approximately 50-60 dB. The volume will be continuously monitored using a sound level meter and adjusted as needed. The music will stop once the airway is secured by the attending anesthetist (i.e. following endotracheal intubation or placement of a laryngeal mask). Music will resume after the surgery is completed, the bandage (if required) has been applied, and the administration of anesthetic medication has ceased. Music will be paused again after anesthesia emergence as the patient leaves the operating room.
  Interventions: Other: Music
- Control group (No Intervention): The control group will not receive music during anesthesia induction or emergence. However, the State Trait Anxiety Inventory (STAI) will be administered preoperatively as well as the State Anxiety Inventory (SAI) portion of the STAI postoperatively.

INTERVENTIONS:
Other: Music — Music as per patient choice
  Arms: Music group

SUMMARY:
Perioperative anxiety remains a prevalent and significant concern for patients undergoing surgery, with substantial impacts on postoperative pain perception, patient satisfaction and recovery. Historically, anxiolytics (e.g. benzodiazepines) were often routinely administered preoperatively in this context, accepting the potential negative side effects of pharmacotherapy. In recent literature, there is an increasing focus on alternative, non-pharmacological methods for anxiety reduction, such as music, music therapy, virtual reality, and hypnosis.

Music can represent an effective and cost-efficient option to reduce perioperative anxiety and stress. Most randomized controlled trials on this topic (music group vs. non-music group) have been conducted in pediatric patient populations, often showing significant results (i.e. significantly less anxiety in the music group, measured using standardized scales or inventories). In adult patient populations, considerably fewer randomized controlled trials with music interventions for perioperative anxiety reduction have been conducted so far.

This study aims to evaluate the role of music during anesthesia induction and emergence for perioperative anxiety reduction in a randomized controlled trial. Patients will be randomized preoperatively into either the intervention group (50 patients, music) or the control group (50 patients, no music), and a baseline level of preoperative anxiety will be assessed using the State-Trait Anxiety Inventory (STAI). In the intervention group, music of the patient's choice will be played starting from their arrival in the operating room during anesthesia induction, and again after the end of surgery during emergence from anesthesia. Afterwards, the effects of the music intervention on the patients' subjective well-being will be assessed in the intervention group postoperatively before discharge from the recovery room using four specific questions. In both groups, the State Anxiety Inventory (SAI) portion of the STAI will also be administered and the results compared.

In addition, the NASA Task Load Index will be administered to the attending anesthesiologists in both groups to evaluate whether the subjective workload of the anesthesiologists changes as a result of the music intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Elective ophthalmological surgery under general anesthesia (e.g. strabismus surgery, cataract surgery or other lens surgery, glaucoma surgery, keratoplasty or other corneal transplantation, vitrectomy or other retinal surgery, lacrimal duct surgery)
* Age: 18-70 years
* ASA score I-II (American Society of Anesthesiologists)

Exclusion Criteria:

* Pre-existing psychiatric disorder (e.g. anxiety disorder, PTSD, depression)
* Chronic pain patients
* Language barrier
* Anticipated difficult airway
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Impact of listening to self-selected music during anesthesia induction and emergence on patient well-being | Postoperatively before discharge from the post-anesthesia care unit (PACU)
  The primary objective of this randomized controlled trial is to assess the impact of listening to self-selected music during anesthesia induction and emergence on patient well-being, as measured by four specific questions:
  1. I enjoyed listening to the music I chose, during the anesthesia induction and emergence.
  2. Listening to the music I chose, during anesthesia induction and emergence had an anxiety relieving effect.
  3. Listening to the music I chose, during anesthesia induction and emergence had a stress-relieving effect.
  4. The next time I have a general anesthesia, I would like to listen to self-selected music during anesthesia induction and emergence.
  These questions will be answered using a Likert scale (strongly disagree - disagreee - neither agree nor disagree - agree - strongly agree).

SECONDARY OUTCOMES:
Sex-specific differences regarding the primary objective | Postoperatively before discharge from the post-anesthesia care unit (PACU)
State Trait Anxiety Inventory (STAI) | Pre- and postoperatively
  State Anxiety Inventory (SAI): pre- and postoperatively Trait Anxiety Inventory (TAI): preoperatively
NASA Task Load Index (attending anesthesiologist) | After anesthesia induction + after handover to the post-anesthesia care unit (PACU) team
  The NASA Task Load Index will be completed twice by the attending anesthesiologist in the presence of the study team: once after anesthesia induction, once patient stability and adequate anesthesia are confirmed, and again after anesthesia delivery, once the patient is stable in the post-anesthesia care unit (PACU) and all relevant information has been relayed to the PACU team.
Attempts at airway management | After anesthesia induction
  Intubation attempts Attempts to place a laryngeal mask
Adverse events | During surgery
  Including but not limited to:
  Difficult intubation > 3 attempts Respiratory complications (e.g. bronchospasm, laryngospasm) Hemodynamic complications (severe hypotension (MAP >50 for more than 5 minutes), severe bradycardia (heart rate < 40)) Cardiac arrest
Postoperative pain in the post-anesthesia care unit (PACU) | During the stay in the post-anesthesia care unit (PACU)
  Opioid equivalents Non-opioid analgetic medication

CONTACTS AND LOCATIONS:
Overall Officials: Marion Wiegele, Priv.-Doz. DDr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No